CLINICAL TRIAL: NCT05275595
Title: A Descriptive Study of COVID-19 Among Children With Chronic Renal Diseases in Qatar
Brief Title: COVID-19 Among Children With Chronic Renal Diseases in Qatar
Acronym: CCCRDQ
Status: Completed | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-22-052
Record Dates: First submitted 2022-03-08; First posted 2022-03-11 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Diseases; COVID-19 Infection; Acute Kidney Injury; Chronic Renal Failure in Children; COVID-19 Pandemic
MeSH Terms: conditions — Renal Insufficiency, Chronic; COVID-19; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chronic renal disease with covid: all patients who have chronic kidney disease with COVID-19 infection
  Interventions: Other: Medical records review
- chronic renal disease without covid: all patients who have chronic kidney disease without COVID-19 infection
  Interventions: Other: Medical records review

INTERVENTIONS:
Other: Medical records review — Data on clinical and laboratory findings are reviewed from medical records for details of underlying disease, severity of COVID-19 and associated complications, testing methods for SARS-CoV-2 virus and duration of RT-PCR positivity, therapy received, and duration of hospital stay. Underlying CKD was categorized as nephrotic syndrome, other kidney diseases with CKD stage 1-5. In patients with nephrotic syndrome, the presence of nephrotic-range proteinuria at evaluation at onset, relapse or following non-response to immunosuppression, was considered as 'relapse'.
  The Patients will be followed up until discharge, death or 4weeks after diagnosis of COVID-19, whichever was earlier, until 20 January.
  Groups: chronic renal disease with covid
Other: Medical records review — Data on clinical and laboratory findings are reviewed from medical records for details of underlying disease, associated complications, therapy received, and duration of hospital stay. Underlying CKD was categorized as nephrotic syndrome, other kidney diseases with CKD stage 1-5.
  Groups: chronic renal disease without covid

SUMMARY:
Coronavirus disease 2019 is a novel viral disease caused by the Severe Acute Respiratory Syndrome Coronavirus 2 virus. The original cases occurred in Wuhan, China, in December 2019 and rapidly spread to other areas worldwide, constituting a pandemic with unimaginable health and economic consequences. the World Health Organization elevated the disease to the category of a pandemic on March 11, 2020.

In children, the reported mortality rates were far below 1%, while in people above the age of 70 years it was above 5% or higher. So, in this retrospective study, the investigators describe the clinical features and outcomes of children with chronic kidney diseases who were diagnosed with Severe Acute Respiratory Syndrome Coronavirus 2 infection at pediatric centers in Doha from 1st March 2020 till January 20th, 2022. This review looks into the literature on pediatric patients with chronic kidney diseases to verify whether they were more prone to developing more severe symptoms when diagnosed with Coronavirus disease 2019 compared to children without chronic kidney diseases and adults with chronic kidney diseases, and the Prevalence of COVID-19 infection between patients with chronic kidney diseases, and the role of COVID-19 infection in increasing the relapses and deterioration of chronic kidney diseases.

DETAILED DESCRIPTION:
In this retrospective study investigators will include all children and adolescents (≤ 18 years old) with pre-existing CKD and laboratory-confirmed SARS-CoV-2 infection who were treated at Hamad General Hospital, in Doha, Qatar during this pandemic using the electronic medical records from 1st March 2020 till January 20th, 2022. Indications for testing patients for SARS CoV-2 infection included:

* Clinical features suggestive of COVID-19 (fever, cough, dyspnea, rhinorrhea, sore throat, diarrhea, myalgia, anosmia, or ageusia).
* Close contact (within 6-ft of an infected person for 15 min or longer) within an individual diagnosed with SARS-CoV-2 infection.
* Admission for management of the underlying disease. Testing for SARS-CoV-2 infection was performed on nasal and oropharyngeal swabs using reverse transcriptase polymerase chain reaction (RT-PCR) or rapid antigen test.

Indications for hospital admission were:

* symptomatic infection, particularly in an immunosuppressed host.
* management of the underlying illness.
* inability to ensure home isolation. Data on clinical and laboratory findings are reviewed from medical records for details of underlying disease, the severity of COVID-19 and associated complications, testing methods for SARS-CoV-2 virus and duration of RT-PCR positivity, therapy received, and duration of hospital stay. Underlying CKD was categorized as nephrotic syndrome, other kidney diseases with CKD stage 1-5. In patients with nephrotic syndrome, the presence of nephrotic-range proteinuria at evaluation at onset, relapse, or following non-response to immunosuppression, was considered as 'relapse'.

The Patients will be followed up until discharge, death, or 4weeks after diagnosis of COVID-19, whichever was earlier, until 20 January. Hypertension was defined using standard guidelines. The estimated glomerular filtration rate (eGFR) was calculated using the modified Schwartz formula.

Investigators will look for the clinical manifestations, radiological and laboratory findings, severity of COVID-19 infection, prevalence and difference between waves of the pandemic, median age, gender, and ethnic background. Underlying illness, renal treatment, reinfection, correlation with vaccination.

Participants are divided into three groups; first wave, second wave, and third wave

ELIGIBILITY:
Inclusion Criteria:

* All children and adolescents (≤ 18 years old).
* who have underlying kidney disease.
* laboratory-confirmed SARS-CoV-2 infection.

Exclusion Criteria:

* Patients with SARS-CoV-2 infection who developed AKI during the hospital stay but lacked evidence of pre-existing kidney disease.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This retrospective review of electronic medical records from the Pediatric nephrology division, Pediatrics division, Hamad General hospital in Doha, Qatar, will include all children and adolescents (≤ 18 years old) with pre-existing CKD and laboratory-confirmed SARS-CoV-2 infection between March 2020, to 20 January 2022.
  Approximately 100 eligible records will be reviewed. Data collection will be done by the investigators for all participants.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The relationship between chronic kidney disease and COVID-19 infection in children | 2 year
  There is an increased predisposition to COVID-19 infection in patients with CKD due to illness or treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alhandi Omar Helal, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar